CLINICAL TRIAL: NCT00680472
Title: Protocol HKT-500-US08: A Randomized, Multicenter, Double-blind, Placebo-controlled, Two-week Study to Assess the Efficacy and Safety of HKT-500 in Subjects With Acute Shoulder Pain
Brief Title: HKT-500 in Adult Patients With Shoulder Pain
Acronym: Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hisamitsu Pharmaceutical Co., Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HKT-500-US08
Record Dates: First submitted 2008-05-16; First posted 2008-05-20 (Estimated); Last update posted 2015-06-04 (Estimated); Status verified 2015-05

CONDITIONS: Pain
Keywords: Shoulder pain; Pain; Ketoprofen; Topical Patch
MeSH Terms: conditions — Pain; Shoulder Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A,1 HKT-500 Ketoprofen Topical Patch (Active Comparator): A Randomized, Multicenter, Double-Blind, Placebo-Controlled, Two-Week Study to Assess the Efficacy and Safety of HKT-500 in Subjects with Acute Shoulder Pain
  Interventions: Drug: HKT-500 Ketoprofen Topical Patch
- A,2 Placebo Patch (Placebo Comparator): Treatment with placebo patch
  Interventions: Other: Placebo Patch

INTERVENTIONS:
Drug: HKT-500 Ketoprofen Topical Patch — HKT-500 Ketoprofen Topical Patch
  Other Names: Ketoprofen Topical Patch
  Arms: A,1 HKT-500 Ketoprofen Topical Patch
Other: Placebo Patch — Treatment with Placebo Patch
  Other Names: Sham treatment
  Arms: A,2 Placebo Patch

SUMMARY:
The objective of this study is to determine the efficacy of HKT-500 in subjects with acute shoulder pain

DETAILED DESCRIPTION:
Randomized, double-blind, placebo-controlled, multicenter study in men and women 18 years of age or greater who have acute shoulder pain requiring analgesic treatment daily for at least 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

* The subject has unilateral acute shoulder pain.

Exclusion Criteria:

* The subject is a women of childbearing potential who has a positive urine pregnancy test, or who is lactating, or who is not surgically sterile (by tubal ligation or hysterectomy), or at least 2 years postmenopausal, and has not practiced an acceptable form of birth control (defined as the use of an intrauterine device with spermicide, a barrier method with spermicide, condoms with spermicide, subdermal implant, oral contraceptives, or abstinence) for at least 2 months prior to Visit 1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 368 (Actual)
Dates: Start 2008-04; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Pain Assessment | 2 Weeks

SECONDARY OUTCOMES:
Safety Assessment | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kenichi Furuta, Study Director — Hisamitsu Pharmaceutical Co., Inc.
Locations (33):
- United States (33):
  - Hisamitsu Investigator Site, Birmingham, Alabama
  - Hisamitsu Investigator Site, Tempe, Arizona
  - Hisamitsu Investigator Site, Fullerton, California
  - Hisamitsu Investigator Site, Denver, Colorado
  - Hisamitsu Investigator Site, Washington D.C., District of Columbia
  - Hisamitsu Investigator Site, Bradenton, Florida
  - Hisamitsu Investigator Site, Chiefland, Florida
  - Hisamitsu Investigator Site, DeLand, Florida
  - Hisamitsu Investigator Site, Delray Beach, Florida
  - Hisamitsu Investigator Site, Dunedin, Florida
  - Hisamitsu Investigator Site, Longwood, Florida
  - Hisamitsu Investigator Site, Oldsmar, Florida
  - Hisamitsu Pharmaceutical Co., Inc., Orange City, Florida
  - Hisamitsu Investigator Site, Plantation, Florida
  - Hisamitsu Investigator Site, Tampa, Florida
  - Hisamitsu Investigator Site, Blue Ridge, Georgia
  - Hisamitsu Investigator Site, Boise, Idaho
  - Hisamitsu Investigator Site, Wichita, Kansas
  - Hisamitsu Investigator Site, Paducah, Kentucky
  - Hisamitsu Investigator Site, Bowie, Maryland
  - Hisamitsu Investigator Site, Kalamazoo, Michigan
  - Hisamitsu Investigator Site, Bridgewater, New Jersey
  - Hisamitsu Investigator Site, Cary, North Carolina
  - HIsamitsu Pharmaceutical Co., Inc., Durham, North Carolina
  - Hisamitsu Investigator Site, Raleigh, North Carolina
  - Hisamitsu Investigator Site, Fargo, North Dakota
  - HIsamitsu Pharmaceutical Co., Inc., Perrysburg, Ohio
  - Hisamitsu Investigator Site, Toledo, Ohio
  - Hisamitsu Investigator Site, Zanesville, Ohio
  - Hisamitsu Investigator Site, New Tazewell, Tennessee
  - Hisamitsu Investigator Site, Bryan, Texas
  - Hisamitsu Investigator Site, San Antonio, Texas
  - Hisamitsu Investigator Site, Newport News, Virginia